CLINICAL TRIAL: NCT04094584
Title: Feasibility of Emergency Department Initiated Extended-Release Naltrexone and Case Management Services for the Treatment of Alcohol Use Disorder
Brief Title: Emergency Department Initiated Extended-Release Naltrexone and Case Management for the Treatment of Alcohol Use Disorder
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: 12 month follow up data not collected due to pandemic disruptions
Sponsor: University of California, San Francisco (Other)
Collaborators: Carestar Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-26090
Record Dates: First submitted 2019-09-17; First posted 2019-09-19 (Actual); Results first posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-05

CONDITIONS: Alcohol Use Disorder; Substance Use; Alcohol Abuse or Dependence
Keywords: Emergency Department; Naltrexone
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders; Emergencies | interventions — vivitrol; Case Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Multimodal Intervention (Experimental): The intervention is multimodal and consists of:
  1. Intramuscular injections of 380mg extended-release Naltrexone, given once monthly for 3 months.
  2. Case Management services
  Interventions: Drug: Vivitrol (Extended Release Naltrexone)

INTERVENTIONS:
Drug: Vivitrol (Extended Release Naltrexone) — Monthly Injections of 380mg Extended-Release Naltrexone, case management services as needed tailored to the individual participant
  Other Names: Case Management; SBIRT

SUMMARY:
This is a phase 4, open-label, feasibility study of extended release naltrexone (Vivitrol, Alkermes Pharmaceutical) and case management for treatment of alcohol use disorders in the ED.

Excess alcohol use is a major cause of morbidity and mortality and contributes to a large number of emergency department (ED) visits. The rate of alcohol-related ED visits is increasing, and there is evidence that this increase may be driven by a subset of patients who frequently visit the ED due to an underlying alcohol use disorder (AUD). The proposed study will assess the feasibility of implementing a multimodal treatment for AUD in the emergency department for 25 patients with AUD. The rationale for including each component of the multimodal treatment is outlined below.

Pharmacotherapy is recommended as the standard of care for alcohol use disorders. Of the four drugs approved by the FDA for treatment of alcohol use disorder, extended release naltrexone has been found to be superior at reducing healthcare utilization, increasing detoxification facility use, and reducing total cost. Fewer than 1 in 4 patients with AUD currently receives treatment with an FDA approved agent and use of these drugs in EDs is virtually non-existent.

ED patients with alcohol use disorders frequently suffer from multiple medical, mental health, and social problems that influence their health. Providing such patients with case management services has shown promise in improving health related outcomes while curbing ED utilization and healthcare costs.

Regardless of comorbidity, limited access to substance use and mental health services is a significant barrier to receiving treatment, and large disparities exist in access based on income level. Facilitated referrals, where a healthcare worker communicates with the patient and service providers and assists the patient with obtaining follow up, have been used effectively to improve access to specialty care after ED discharge. Case managers are familiar with community treatment resources and are well versed in providing facilitated referrals.

The primary hypothesis is that implementing this multimodal treatment will be feasible in an ED setting and will reduce alcohol use. Feasibility measures (recruitment, retention, continuation of treatment after the trial) are the primary outcomes. The intent of the intervention is to change drinking behavior in a way that benefits participants' health and quality of life. As such, we will conduct a limited efficacy assessment. Treatment efficacy will be assessed by comparing alcohol consumption, quality of life, and life consequences related to alcohol use before and after the intervention.

The primary efficacy outcome is change in total alcohol consumption measured by a 2 week timeline follow back. Change from baseline will be assessed after the 3 month intervention period, and at the conclusion of the study follow up period for all outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Active alcohol use by self-report
* Known alcohol use disorder or suspected alcohol use disorder and Alcohol Use Disorders Identification Test (AUDIT) score ≥ 8 or AUDIT-C score > 4, or frequent emergency department visits and hazardous drinking defined as: At least 3 emergency department visits in the past 12 months, including the index visit, and Alcohol Use Disorders Identification Test (AUDIT) score ≥ 8 or AUDIT-C score > 4

Exclusion Criteria:

* Opioid use: currently receiving opioid analgesics, self-report of opioid use in past 7 days, current physiologic opioid dependence, patients in acute opioid withdrawal, urine toxicology screen positive for opiates including fentanyl
* History of hypersensitivity to naltrexone, polylactide-co-glycolide (PLG), carboxymethylcellulose, or any other components of the diluent
* Liver function tests (AST, ALT) > 5x upper limit of normal or known cirrhosis
* Platelets less than 100,000 per cubic mm
* Acute condition at the time of enrollment that necessitates medical therapy with opioids
* Pregnant
* Incarcerated

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2020-08-14 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Raven, MD, Principal Investigator — University of California, San Francisco; Charles E Murphy IV, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Murphy CE 4th, Coralic Z, Wang RC, Montoy JCC, Ramirez B, Raven MC. Extended-Release Naltrexone and Case Management for Treatment of Alcohol Use Disorder in the Emergency Department. Ann Emerg Med. 2023 Apr;81(4):440-449. doi: 10.1016/j.annemergmed.2022.08.453. Epub 2022 Oct 31. PMID 36328851

RESULTS

PARTICIPANT FLOW:
Groups:
- Multimodal Intervention: The intervention is multimodal and consists of:
  1. Intramuscular injections of 380mg extended-release Naltrexone, given once monthly for 3 months.
  2. Case Management services
  Extended Release Naltrexone: Monthly Injections of 380mg Extended-Release Naltrexone, case management services as needed tailored to the individual participant
Period: Overall Study
Arm/Group | Multimodal Intervention
Started | 179
Screened for Eligibility (Screened for eligibility based on pre-screening result of being interested and willing to undergo screened) | 55
Enrolled and Received First Injection | 32
Completed | 23
Not Completed | 156
Not completed — No interest in study | 88
Not completed — Unwilling to undergo screening tests | 36
Not completed — Liver disease (enzymes >5 times upper limit of cirrhosis) | 8
Not completed — Opioid use | 7
Not completed — Need for major surgery in study period | 4
Not completed — eligible but declined enrollment | 4
Not completed — Chose to stop injections after week 4 but continued case management and provided complete data | 2
Not completed — Missed study visits resulting. in incomplete data but sufficient for a pre-post comparison | 2
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Multimodal Intervention
Number analyzed (Participants) | 32
Age, Continuous [Median (Full Range); unit: years] | 43 [28 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Demographic characteristics:: White | 23
  Demographic characteristics:: Asian or Pacific Islander | 2
  Demographic characteristics:: Native American | 1
  Demographic characteristics:: LatinX | 6
Annual income [Median (Inter-Quartile Range); unit: U.S. Dollars/ year] | 30,000 [10,000 to 70,000]
Education [Median (Full Range); unit: years] — Highest Grade achieved
  years | 14 [8 to 20]
Employed [Count of Participants; unit: Participants] | 21
Stable housing [Count of Participants; unit: Participants] | 21
Comorbid serious mental illness [Count of Participants; unit: Participants] | 8
Tobacco use [Count of Participants; unit: Participants] | 20
Any comorbid substance use [Count of Participants; unit: Participants] | 16
Amphetamines [Count of Participants; unit: Participants] — comorbid use
  Participants | 7
Cocaine [Count of Participants; unit: Participants] — comorbid use
  Participants | 2
Cannabis [Count of Participants; unit: Participants] — comorbid use
  Participants | 12
Alcohol Use Disorder Identification Test (AUDIT) score [Median (Inter-Quartile Range); unit: units on a scale] — alcohol use disorder identification test consumption score, range 0-12, score > 4 consistent with alcohol misuse and possible liver damage
  units on a scale | 11 [9 to 12]
Daily alcohol consumption over the past 14 days [Median (Inter-Quartile Range); unit: drinks per day] — 1 drink contains 14 grams of ethyl alcohol
  drinks per day | 7.6 [4.8 to 13.2]
WHO drinking risk level [Median (Inter-Quartile Range); unit: units on a scale] — Risk levels for health consequences due to alcohol use: 4 Very High, 3 High, 2 Moderate, 1 Low
  units on a scale | 4 [3 to 4]
Short Inventory of Problems Score (SIP-2R) [Median (Inter-Quartile Range); unit: units on a scale] — Possible score 0-45 with higher scores indicative of more alcohol-related problems. Scores 30-45 and 23-29 indicate "Very High" and "High" levels of alcohol related problems
  units on a scale | 26 [15 to 31]
Kemp Quality of Life Scale Score [Mean (Standard Deviation); unit: units on a scale] — Score range 1-7 with high scores indicating better quality of life
  units on a scale | 3.6 (1.7)

OUTCOME MEASURES:

1. Primary Outcome: Participants Retained in Study at 3 Months
Description: Percentage of enrolled participants who attend final study visit at the end of the intervention period
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Groups:
- Multimodal Intervention: The intervention is multimodal and consists of:
  1. Intramuscular injections of 380mg extended-release Naltrexone, given once monthly for 3 months.
  2. Case Management services
  Vivitrol (Extended Release Naltrexone): Monthly Injections of 380mg Extended-Release Naltrexone, case management services as needed tailored to the individual participant
Arm/Group | Multimodal Intervention
Number analyzed (Participants) | 32
Participants | 27

2. Primary Outcome: Retention at 12 Months
Description: Percentage of enrolled participants who complete final study visit at the end of the follow up periods
Time Frame: 12 months
Population: These data were not collected due to COVID-19 pandemic disruptions.
Arm/Group | Multimodal Intervention
Number analyzed (Participants) | 0

3. Primary Outcome: Change in Daily Total Alcohol Consumption From Baseline at 3 Months
Description: Self-reported total daily alcohol consumption at 3 months, compared to baseline
Time Frame: 3 months after enrollment
Measure: Median (95% Confidence Interval); unit: drinks per day
Arm/Group | Multimodal Intervention
Number analyzed (Participants) | 27
drinks per day | -7.5 [-8.6 to -5.9]

4. Primary Outcome: Change in Total Alcohol Consumption at 12 Months
Description: Change in self-reported total daily alcohol consumption from baseline
Time Frame: 12 months after enrollment
Population: These data were not collected due to COVID-19 pandemic disruptions.
Arm/Group | Multimodal Intervention
Number analyzed (Participants) | 0

5. Secondary Outcome: Change in Quality of Life Score at 3 Months
Description: Kemp Quality of Life score at 3 months compared to baseline. Score is 1-7 with higher scores indicating higher quality of life.
Time Frame: 3 months after enrollment
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Multimodal Intervention
Number analyzed (Participants) | 27
score on a scale | 1.2 [0.5 to 1.9]

6. Other Pre Specified Outcome: Substance Use Treatment Utilization
Description: percentage of participants self-reporting engagement in community substance use treatment programs
Time Frame: 12 months
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Recruitment
Description: Percentage of those approached who enroll in the study
Time Frame: 12 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Continued Naltrexone Use After Intervention Period
Description: Percentage of enrolled who self reported continuing treatment with naltrexone through their primary physician after the end of the study intervention period
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Multimodal Intervention
Number analyzed (Participants) | 32
Participants | 22

9. Other Pre Specified Outcome: Change in ED Utilization
Description: Change in the number of emergency department visits determined by electronic medical record review
Time Frame: 12 months before and after enrollment
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Change in WHO Drinking Risk Level
Description: Change in World Health Organization drinking risk level from baseline. Risk levels are scored 1-4 with higher scores indicating more severe health risk from alcohol use
Time Frame: 3 months after enrollment
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Multimodal Intervention
Number analyzed (Participants) | 27
score on a scale | -2 [-3 to 0]

11. Other Pre Specified Outcome: Change in Alcohol Related Life Consequences (Short Inventory of Problems Scale, Version 2R: SIP-2R)
Description: Change in life consequences due to alcohol use from baseline as measured by revised short inventory of problems (score 0-45 with higher scores indicating more severe alcohol related life consequences)
Time Frame: 3 months after enrollment
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Multimodal Intervention
Number analyzed (Participants) | 27
score on a scale | -13 [-19 to -7]

12. Other Pre Specified Outcome: Receipt of All Study Naltrexone Injections
Description: Percentage of participants receiving all 3 scheduled naltrexone injections received
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Multimodal Intervention
Number analyzed (Participants) | 32
Participants | 23

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Multimodal Intervention
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-11): https://cdn.clinicaltrials.gov/large-docs/84/NCT04094584/Prot_SAP_000.pdf